CLINICAL TRIAL: NCT05040347
Title: Neutrophil Extracellular Traps as a Biomarker to Predict Portal Vein Tumor Thrombosis in Patients With Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYWZLL26511
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Neutrophil Extracellular Trap Formation; Portal Vein Tumor Thrombosis
Keywords: Neutrophil Extracellular Trap; Portal Vein Tumor Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PVTT group: The diagnosis of portal vein tumor thrombosis was confirmed by clinical correlation using histologic features taken from liver biopsy as determined by a pathologist,and findings from image studies including ultrasound, computed tomography, and MRI, verified by a radiologist.
  Interventions: Other: test NETs markers
- HCC group: The diagnosis of HCC was confirmed by clinical correlation using histologic features taken from liver biopsy as determined by a pathologist,and findings from image studies including ultrasound, computed tomography, and MRI, verified by a radiologist.
  Interventions: Other: test NETs markers
- control group: The presence of PVTT or HCC was confirmed by medical record review and all the recorded events were confirmed by a radiologist using imaging studies, ultrasound, contrast-enhanced, or MR.
  Interventions: Other: test NETs markers

INTERVENTIONS:
Other: test NETs markers — NETs markers (Myeloperoxidase, Neutrophil elastase, Citrate histone H3) and anti-β2 glycoprotein I were detected in plasma using capture ELISA and specific ELISA kits.

SUMMARY:
The aim of this study was to investigate whether NETs markers can enhance predict portal vein tumor thrombosis in patients with live cirrhosis, so as to establish a novel predictor to guide clinical decision-making.

DETAILED DESCRIPTION:
Eighty-six patients with patients treated at the Affiliated Hospital of Qingdao University (China) from September 2020 to January 2021 were recruited for this study, including 14 patients with portal vein tumor thrombosis, 28 patients without portal vein tumor thrombosis and 44 patients without hepatocellular carcinoma. NETs markers (Myeloperoxidase, Neutrophil elastase, Citrate histone H3), and anti-β2 glycoprotein I were detected in plasma using capture ELISA and specific ELISA kits. T-test was performed to analyze whether there was a statistical difference between the two groups, and regression analysis was performed between NETs markers and tissue factor and anti-β2 glycoprotein I to investigate whether there was a correlation. This study without any intervention measures, will not cause harm.

ELIGIBILITY:
Inclusion Criteria:

（1) Clinical diagnosis of HCC with liver cirhosis (2) Clinical diagnosis of portal vein tumor thrombosis

Exclusion Criteria:

(1) secondary liver malignancy (2)hematologic diseases (3) Bud-Chiah syndrome (4) incomplete data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty-six patients with patients treated at the Affiliated Hospital of Qingdao University (China) from September 2020 to January 2021 were recruited for this study, including 14 patients with portal vein tumor thrombosis, 28 patients without portal vein tumor thrombosis and 44 patients without hepatocellular carcinoma.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Concentration of NETs markers and anti-β2 glycoprotein I | 1 year.
  NETs markers (Myeloperoxidase, Neutrophil elastase, Citrate histone H3) and anti-β2 glycoprotein I were detected in plasma using capture ELISA and specific ELISA kits.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided